CLINICAL TRIAL: NCT04154293
Title: A Randomized, Parallel, Double-Blind, Vehicle Controlled Study to Evaluate the Safety and Efficacy of Two Concentrations of Topical TMB-001 for the Treatment of Congenital Ichthyosis
Brief Title: A Vehicle Controlled Study to Evaluate Safety and Efficacy of Topical TMB-001 for Treatment of Congenital Ichthyosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Timber Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 235-9051-202; 1R01FD006079-01A1 (FDA)
Record Dates: First submitted 2019-11-01; First posted 2019-11-06 (Actual); Results first posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Congenital Ichthyosis
MeSH Terms: conditions — Ichthyosis Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Intervention Model Description: A Randomized, Parallel, Double-Blind, Vehicle-Controlled Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vehicle Ointment (Control) (Placebo Comparator): Topical, BID (Twice daily)
  Interventions: Other: Vehicle
- TMB-001 Ointment, 0.05% (Experimental): Topical, BID ( twice daily)
  Interventions: Drug: Isotretinoin
- TMB-001 Ointment, 0.1% (Experimental): Topical, BID (Twice daily)
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin — Topical Isotretinoin ointment
  Other Names: TMB-001
  Arms: TMB-001 Ointment, 0.05%; TMB-001 Ointment, 0.1%
Other: Vehicle — Topical Vehicle Ointment
  Arms: Vehicle Ointment (Control)

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of two concentrations of topically applied ointment formulation of isotretinoin called TMB-001 (0.05% and 0.1% isotretinoin) in subjects 9 years of age and older for the treatment of congenital ichthyosis (CI), including recessive X-linked ichthyosis (RXLI) and autosomal recessive congenital ichthyosis-lamellar ichthyosis (ARCI-LI) subtypes.

Funding Source FDA-OOPD

DETAILED DESCRIPTION:
This is a randomized, parallel, double-blind, vehicle-controlled study to evaluate the safety and efficacy of two concentrations of topical TMB-001 for the treatment of CI in subjects with either the ARCI-LI or RXLI subtypes. The duration of treatment will be 12 weeks. Each subject will participate in the study for up to 24 weeks (including up to a 90-day Screening period). Eleven study centers from United States of America and Australia participated in this global study. Each subject participated in the study for up to 24 weeks (including up to a 90-day Screening period).

Eligible subjects were randomized (1:1:1) to one of 3 treatment groups:

1. TMB-001, 0.05%, twice daily (bid)
2. TMB-001, 0.1%, bid
3. Vehicle Ointment (Control), 0%, bid

Subjects were evaluated on a monthly basis for safety and efficacy results over the 12- week treatment period. Efficacy was determined in 2 ways:

1. VIIS (or Visual Index of Ichthyosis Severity) "treatment success" (VIIS-50) was defined as ≥ 50% reduction from Baseline for VIIS scaling score for the sum of the scores for 'VIIS body areas' that had a Baseline score ≥ 3). The proportion of subjects achieving VIIS-50 at Visit 6 at Week 12 relative to Baseline was the primary efficacy endpoint and time point used to compare the two active treatments to vehicle.
2. The proportion of subjects achieving IGA (Investigator Global Assessment) treatment success will be the key secondary endpoint. For this endpoint, the IGA score was established as "treatment success" or "treatment failure" where "treatment success" is defined as at least a 2-grade decrease in severity score (for example, severe or score of 4 at baseline to mild or score of 2 at Visit 6) relative to Baseline at Visit 6 at week 12.

The safety analyses conducted were extent of exposure, changes in physical examinations and vital signs, blood and urine testing including urine pregnancy testing as indicated, local skin reactions (including burning/stinging, redness, erosions, and swelling) and other adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, 9 years of age or older at Visit 2 (Baseline)
* Subject has provided written informed consent
* Females of child bearing potential must be surgically sterile or agree to 2 forms of birth control
* Subject has clinical diagnosis of Congenital Ichthyosis with genetic confirmation of subtype
* Subject has between 10% and 90% total BSA affected by Congenital Ichthyosis
* Subject has at least 2 VIIS assessment areas with a scaling score of 3 or greater

Exclusion Criteria:

* Subject has inflammatory skin diseases unrelated to ichthyosis
* Subject has used other prohibited topical treatments in the assessment areas within certain days from baseline
* Subject has used systemic retinoids within12 weeks of baseline
* Subject has untreated secondary infections
* Subject has lesions suspicious for skin cancer or untreated skin cancers

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan M Mendelsohn, MD, Study Director — Timber Pharmaceuticals
Locations (11):
- United States (8):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Stanford University School of Medicine, Palo Alto, California
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Austin Institute for Clinical Research, Inc, Metairie, Louisiana
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Australia (3):
  - Queensland Children's Hospital, Brisbane, Queensland
  - Premier Specialists, The church, Kogarah, Sydney
  - Murdoch Children's Research Institute, RCH, Melbourne, Victoria

REFERENCES:
- [Derived] Marathe K, Teng JMC, Guenthner S, Bunick CG, Kempers S, Eads K, Castelo-Soccio L, Mendelsohn AM, Raiz J, Murrell DF. Topical Isotretinoin (TMB-001) Treatment for 12 Weeks Did Not Result in Clinically Relevant Laboratory Abnormalities in Participants with Congenital Ichthyosis in the Phase 2b CONTROL Study. Dermatol Ther (Heidelb). 2023 Jun;13(6):1255-1264. doi: 10.1007/s13555-023-00923-1. Epub 2023 May 11. PMID 37170057

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle Ointment (Control) | TMB-001 Ointment, 0.05% | TMB-001 Ointment, 0.1%
Started | 12 | 11 | 11
Number Who Received at Least 1 Dose | 12 | 11 | 10
Completed | 10 | 8 | 9
Not Completed | 2 | 3 | 2
Not completed — Withdrawal by Subject | 2 | 3 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one dose of study drug (TMB-001 0.1% or TMB-001 0.05%) or vehicle
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle Ointment (Control) | TMB-001 Ointment, 0.05% | TMB-001 Ointment, 0.1% | Total
Number analyzed (Participants) | 12 | 11 | 10 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (24.6) | 31.9 (18.6) | 34.5 (19.7) | 34.5 (20.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 12
  Male | 8 | 8 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 1 | 6
  Not Hispanic or Latino | 9 | 9 | 9 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 10 | 8 | 8 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 9 | 32
  Australia | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Reduction in Targeted Ichthyosis Severity Using the Visual Index for Ichthyosis Severity Measurement
Description: Number of subjects with Visual Index for Ichthyosis Severity (VIIS) treatment success, defined as 50% or greater decreased in VIIS scaling score
Time Frame: 12 weeks
Population: Intention to treat analysis only on subjects who received at least one dose of study medication; one subject in TMB-001 0.1% arm was randomized but never received study medication due to COVID
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Ointment (Control) | TMB-001 Ointment, 0.05% | TMB-001 Ointment, 0.1%
Number analyzed (Participants) | 12 | 11 | 10
Participants | 4 | 7 | 4

2. Secondary Outcome: Number of Subjects With Reduction in Overall Ichthyosis Severity as Measured With Investigator Global Assessment
Description: Number of subjects with Investigator Global Assessment decrease in disease severity by at least 2 grades
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Ointment (Control) | TMB-001 Ointment, 0.05% | TMB-001 Ointment, 0.1%
Number analyzed (Participants) | 12 | 11 | 10
Participants | 1 | 6 | 4

3. Secondary Outcome: Change in I-NRS (Itch-Numeric Rating Scale) From Baseline at Week 12
Description: Mean numeric Change from baseline in Itch-Numeric Rating Scale (I-NRS) at Week 12 for entire population. I-NRS is an 11-point visual analogue scale scored based upon 0 being no itch and 10 being worst itch imaginable. Subjects were asked to grade their itch on such a scale at each visit where I-NRS was administered. A 4-point change from baseline is considered clinically significant
Time Frame: 12 weeks
Population: Intention to treat analysis based upon available data collected. Data imputation was not performed for I-NRS but only for primary endpoint as above
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle Ointment (Control) | TMB-001 Ointment, 0.05% | TMB-001 Ointment, 0.1%
Number analyzed (Participants) | 10 | 9 | 9
units on a scale | -1.7 (2.54) | -1.9 (5.3) | 1.1 (2.64)

4. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 12
Description: Change from Baseline in Dermatology Life Quality Index (DLQI) at Week 12 in all adult subjects.
  The DLQI is validated in all subjects over age 16 years and is a 10-question questionnaire which requests information on how the dermatological condition affects different aspects of their life. Each question is scored on a 0-3 scale (0=no impact, 3=major impact) for a total possible maximal score of 30. Scores over 11 in adults are considered to indicate moderate impairment of quality of life due to the skin disease. A 4-point improvement from baseline is considered clinically significant
Time Frame: 12 weeks
Population: Intention to treat analysis based upon available data collected. Data imputation was not performed for DLQI but only for primary endpoint as above
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle Ointment (Control) | TMB-001 Ointment, 0.05% | TMB-001 Ointment, 0.1%
Number analyzed (Participants) | 8 | 6 | 7
units on a scale | -3.4 (4.72) | -3.2 (9.28) | -1.3 (3.95)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: follows clinicaltrials.gov definitions. Analysis of adverse events, serious adverse events and other adverse events only on subjects who received at least one dose of study medication; one subject in TMB-001 0.1% arm was randomized but never received study medication due to COVID
Arm/Group | Vehicle Ointment (Control) | TMB-001 Ointment, 0.05% | TMB-001 Ointment, 0.1%
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 3/12 | 9/11 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Ointment (Control) (N=12) | TMB-001 Ointment, 0.05% (N=11) | TMB-001 Ointment, 0.1% (N=10)
palipations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
application site dermatitis (General disorders) | 0 (0) | 3 (6) | 1 (2)
application site discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
application site erosion (General disorders) | 0 (0) | 2 (3) | 1 (2)
application site erythema (General disorders) | 0 (0) | 3 (4) | 4 (5)
application site hypersensitivity (General disorders) | 0 (0) | 0 (0) | 2 (2)
application site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
application site edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
application site pain (General disorders) | 0 (0) | 2 (3) | 3 (6)
application site pruritis (General disorders) | 0 (0) | 3 (5) | 4 (5)
application site rash (General disorders) | 0 (0) | 1 (1) | 0 (0)
application site warmth (General disorders) | 1 (1) | 0 (0) | 0 (0)
acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
application site folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
application site pustules (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
folliculitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
small sample size. study not powered for statistical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT04154293/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04154293/SAP_001.pdf